CLINICAL TRIAL: NCT00288899
Title: Benefits of 'Repeat Back' Protocols Within A Computer-Based Informed Consent Program
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IAF 05-308
Record Dates: First submitted 2006-02-06; First posted 2006-02-08 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Surgery; Cholecystectomy, Laparoscopic; Prostatectomy; Arthroplasty, Replacement, Hip; Endarterectomy, Carotid
Keywords: Informed Consent; Medical Record Systems, computerized; Comprehension; Anxiety; Personal Satisfactin
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Other): standard VA surgical iMedConsent process
  Interventions: Other: standard surgical iMedConsent process
- Arm 2 (Experimental): enhanced version of VA surgical iMedConsent process (repeat-back)
  Interventions: Other: Enhanced surgical iMedConsent process (with "repeat back")

INTERVENTIONS:
Other: Enhanced surgical iMedConsent process (with "repeat back") — Consent process engages patient in discussion about why they are having procedure, risks, benefits, alternatives. Then provider asks patient to "repeat back"what they understand.
  Arms: Arm 2
Other: standard surgical iMedConsent process — Patients are consented in standard VA consent process, where are not necessarily asked to repeat back and no discussion is necessarily documented.
  Arms: Arm 1

SUMMARY:
This is a VA Merit Review Study involving 7 VA medical centers participating in a parallel group randomized trial comparing "repeat back" versus standard electronic consent for 4 common elective surgical procedures (total hip arthroplasty, carotid endarterectomy, laparoscopic cholecystectomy, and radical prostatectomy). Baseline covariates include health status (SF-12), reading ability (REALM), and demographics. Primary outcomes are patient comprehension of the informed consent, patient satisfaction with the informed consent and decision making processes, patient satisfaction with care, anxiety (STAI), and provider assessment of the "repeat back" process. In addition, we are electronically capturing data detailing time spent in each phase of the consent process including "repeat back".

DETAILED DESCRIPTION:
Background: Informed consent for surgical procedures is critical to patient care in the VA and in other health care settings. Many studies document limitations in current methods of obtaining informed consent. These limitations include poor patient comprehension, inadequate time for discussion, poor documentation of consent, and heightening of patient anxiety regarding surgery. In hopes of addressing these shortcomings, both the NQF and AHRQ have recommended that "repeat back" protocols be added to informed consent methodologies. The VA has opted to address the informed consent issue by computerization of the informed consent process utilizing the iMedConsent program. This latter program is fully integrated with the computerized patient record system (CPRS), includes extensive patient education materials, standardizes risk information and guides the clinician through the consent process. The iMedConsent program is being disseminated via an ongoing national rollout. Despite its apparent advantages, the current iMedConsent platform does not incorporate any methodology to support "repeat back". Dialog Medical, the iMedConsent vendor, has recently developed a new module that can enhance the current version of the program by supporting "repeat back" protocols.

Objectives: We hypothesize that use of the enhanced iMedConsent program (with "repeat back") will improve the surgical patient's comprehension about the surgical technique, treatment alternatives, and risks and benefits of the proposed surgery in comparison with the standard iMedConsent program. We believe that this enhanced program will also lead to better patient satisfaction with the consent process, decision making and the health care received, less anxiety about the operation, and that this program will be acceptable to surgical providers and might lead to better clinical outcomes.

Methods: To address these hypotheses we are conducting a multi-site (7 VA Medical Centers) randomized trial comparing the use of the "standard" and "enhanced" iMedConsent program. We will enroll 600 subjects who are scheduled for elective surgery. Subjects will be individually randomized to the standard or enhanced versions of the iMedConsent program. The surgical procedures to be studied include carotid endarterectomy, total hip arthroplasty, radical prostatectomy and laparoscopic cholecystectomy. The study will be linked to the National Surgical Quality Improvement Program data which will provide baseline data on patient characteristics, intraoperative variables (e.g. operation type, time, anesthesia method, etc.), and the data on 30 day surgical outcomes. We will assess endpoints including patient comprehension, patient satisfaction with the consent process, patient anxiety, providers' acceptance of the informed consent process, and patient satisfaction with health care and with decision making using validated self-report survey instruments.

Findings: We are currently in the final phase of data analysis. The final study report will be submitted within the next several weeks to HSR&D.

Status: Study recruitment and enrollment began in August 2006 and ended June 30, 2008. 575 study subjects were randomized, with 502 study subjects completing the study. 214 surgical providers participated and 192 completed provider questionnaires. We continue with final data analysis phase of the study. Manuscripts are being written, with final HSR&D report due within the next several weeks.

Impact: The results of this study will have important implications for improving the consent process within the VA and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Veterans who are scheduled for one of the four elective surgical procedures;
* who give informed consent to participate in the study;
* and who are also part of the NSQIP.

Exclusion Criteria:

* Inability to give informed consent;
* requirement for surrogate consent;
* non-elective surgery;
* requirement for more than one elective surgery;
* refusal to participate;
* inability to communicate in English;
* severe visual problems;
* severe psychiatric illness;
* ongoing substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 575 (Actual)
Dates: Start 2006-08-07 (Actual); Primary Completion 2009-03-31 (Actual); Study Completion 2009-03-31 (Actual)

PRIMARY OUTCOMES:
Patient comprehension; Patient satisfaction; Patient anxiety; Patient compliance; Provider acceptance | 45 days

SECONDARY OUTCOMES:
Risk-adjusted surgical outcomes | Surgical outcome data is collected by VA NSQIP program within 45 days of each surgical procedure. This data will be linked with study data at end of study enrollment, during the data analysis phase.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron S Fink, MD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (7):
- United States (7):
  - VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

REFERENCES:
- [Result] Kaafarani HM, Itani KM. Classification versus valuation and grading of surgical complications. J Am Coll Surg. 2009 Aug;209(2):290-1; author reply 291-2. doi: 10.1016/j.jamcollsurg.2009.05.020. No abstract available. PMID 19632618
- [Result] Itani KM. Let us not forget the Association of VA Surgeons (AVAS). Surgery. 2009 Sep;146(3):525; author reply 525-6. doi: 10.1016/j.surg.2008.11.013. No abstract available. PMID 19715815
- [Result] Itani KM, Kim L. Mechanical bowel preparation or not for elective colorectal surgery. Surg Infect (Larchmt). 2008 Dec;9(6):563-5. doi: 10.1089/sur.2008.9957. PMID 19216667
- [Result] Itani KM, Akhras KS, Stellhorn R, Quintana A, Budd D, Merchant S. Outcomes associated with initial versus later vancomycin use in patients with complicated skin and skin-structure infections. Pharmacoeconomics. 2009;27(5):421-30. doi: 10.2165/00019053-200927050-00006. PMID 19586079
- [Result] Fink AS, Prochazka AV, Henderson WG, Bartenfeld D, Nyirenda C, Webb A, Berger DH, Itani K, Whitehill T, Edwards J, Wilson M, Karsonovich C, Parmelee P. Predictors of comprehension during surgical informed consent. J Am Coll Surg. 2010 Jun;210(6):919-26. doi: 10.1016/j.jamcollsurg.2010.02.049. PMID 20510800
- [Result] Fink AS, Prochazka AV, Henderson WG, Bartenfeld D, Nyirenda C, Webb A, Berger DH, Itani K, Whitehill T, Edwards J, Wilson M, Karsonovich C, Parmelee P. Enhancement of surgical informed consent by addition of repeat back: a multicenter, randomized controlled clinical trial. Ann Surg. 2010 Jul;252(1):27-36. doi: 10.1097/SLA.0b013e3181e3ec61. PMID 20562609
- [Result] Rosen AK, Loveland SA, Romano PS, Itani KM, Silber JH, Even-Shoshan OO, Halenar MJ, Teng Y, Zhu J, Volpp KG. Effects of resident duty hour reform on surgical and procedural patient safety indicators among hospitalized Veterans Health Administration and Medicare patients. Med Care. 2009 Jul;47(7):723-31. doi: 10.1097/MLR.0b013e31819a588f. PMID 19536029
- [Result] Volpp KG, Rosen AK, Rosenbaum PR, Romano PS, Itani KM, Bellini L, Even-Shoshan O, Cen L, Wang Y, Halenar MJ, Silber JH. Did duty hour reform lead to better outcomes among the highest risk patients? J Gen Intern Med. 2009 Oct;24(10):1149-55. doi: 10.1007/s11606-009-1011-z. Epub 2009 May 20. PMID 19455368
- [Derived] Prochazka AV, Fink AS, Bartenfeld D, Henderson WG, Nyirenda C, Webb A, Berger DH, Itani K, Whitehill T, Edwards J, Wilson M, Karsonovich C, Parmelee P. Patient perceptions of surgical informed consent: is repeat back helpful or harmful? J Patient Saf. 2014 Sep;10(3):140-5. doi: 10.1097/PTS.0b013e3182a00317. PMID 24522223